CLINICAL TRIAL: NCT05949762
Title: The Second Affiliated Hospital of Kunming Medical University
Brief Title: Safety and Efficacy of Venetoclax in Combination With Azacitidine and HA Regimen in the Treatment of AML in the Elderly
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ZePing Zhou (Other)
Collaborators: Handan Central Hospital (Other); Taian City Central Hospital (Other); Tianjin People's Hospital (Other); Guizhou Provincial People's Hospital (Other); Second Xiangya Hospital of Central South University (Other); Western War Zone General Hospital (Unknown)
Responsible Party: Sponsor-Investigator, ZePing Zhou, Dr., The Second Affiliated Hospital of Kunming Medical University
Organization: The Second Affiliated Hospital of Kunming Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEN-PJ-KE-2023-157
Record Dates: First submitted 2023-07-10; First posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Venetoclax in Combination With Azacitidine and HA Regimen (Experimental): Details for:
  Venetoclax 200mg d1-10 Azacitidine 100mg/d (or 50-75mg/m2/d), d2-7 Hautriacontin 2mg/m2/d, d3-7 Cytarabine 100mg/m2/d, d3-8 (infusion 24h)
  Interventions: Procedure: Venetoclax in Combination With Azacitidine and HA Regimen

INTERVENTIONS:
Procedure: Venetoclax in Combination With Azacitidine and HA Regimen — Patients diagnosed with primary AML based on morphology, immunophenotyping, and history and meeting the inclusion exclusion criteria were induced with Venetoclax in combination with Azacitidine and HA regimen.
  Details for:
  Venetoclax 200mg d1-10 Azacitidine 100mg/d (or 50-75mg/m2/d), d2-7 Hautriacontin 2mg/m2/d, d3-7 Cytarabine 100mg/m2/d, d3-8 (infusion 24h)

SUMMARY:
This is a prospective phase II, single-arm clinical study that plans to enroll 45 patients aged 60 years or older with primary AML diagnosed after April 1, 2023.The purpose of this trial is to evaluate the efficacy of Venetoclax in combination with azacitidine and HA regimens in elderly patients aged >60 years with primary acute myeloid leukemia and to provide evidence for optimal selection of clinical treatment regimens.

DETAILED DESCRIPTION:
Patients diagnosed with primary AML according to morphology, immunophenotyping and medical history and meeting the exclusion criteria for enrollment: induction therapy with Venetoclax combined with azacitidine and HA regimen, after induction therapy up to CR, CRi, MLFS, according to ELN prognostic stratification and NCCN and Chinese guidelines for the treatment of adult AML (non-acute promyelocytic leukemia), according to patient risk stratification and treatment For patients with allogeneic hematopoietic stem cell transplantation due to various reasons (financial, physical, and other reasons), the patient will be recommended for transplantation. Patients who are not considered for allogeneic HSCT due to various reasons (financial, physical, donor constraints, etc.) will continue to receive two courses of intensive treatment with Venetoclax combined with a medium-dose Ara-c regimen and three courses of reduced-dose chemotherapy for consolidation. Patients completing intensive consolidation therapy enter maintenance treatment with Venetoclax in combination with azacitidine, danazol and thalidomide. Patients who do not achieve CR, CRi and MLFS with 1 course of induction therapy will be re-induced with the original regimen if they achieve PR. Patients who did not achieve PR on the first induction treatment and did not achieve CR, CRi, and MLFS after two induction treatments were dropped from the group and given salvage therapy. Patients with persistent positive MRD or recurrence during treatment were withdrawn from the group and given salvage therapy.

ELIGIBILITY:
Inclusion Criteria:

1. patients with acute myeloid leukemia other than APL who meet the World Health Organization diagnostic criteria (WHO 2016 criteria);
2. those with AML not otherwise classified under the World Health Organization AML classification except for acute myeloproliferative disorder with myelofibrosis and myeloid sarcoma.
3. Age > 60 years, male or female.
4. Have a score of 0-2 on the Eastern Cooperative Oncology Group Physical Status Scale (ECOG-PS).
5. pass the requirements of the following laboratory test indicators (performed within 7 days prior to treatment): 1) Aspartate aminotransferase (ALT), alanine aminotransferase (AST), and alkaline phosphatase (ALP) ≤ 3 x upper limit of normal (ULN), serum bilirubin ≤ 2 x ULN; serum cardiac enzymes < 2.0 x ULN; serum creatinine ≤ 2.0 x ULN; 2) Cardiac ejection fraction within normal values as determined by cardiac ultrasound (ECHO).
6. Informed consent had to be signed before all specific study procedures were started, and the informed consent was signed by the patient himself/herself or his/her immediate family members; in view of the patient's condition, if the signature of the patient himself/herself was not conducive to the treatment of his/her condition, the informed consent was signed by his/her legal guardian or the patient's immediate family members.

Exclusion Criteria:

1、Treated patients (is defined as having received induction chemotherapy in the past, regardless of the efficacy).

2, Concurrent malignant tumors of other organs (those requiring treatment). 3, Patients participating in the trial must use contraception during the trial treatment and within 3 years after completion of treatment.

4, Significantly abnormal liver and kidney function beyond the enrollment criteria.

5. Active heart disease, defined as one or more of the following:

1. History of uncontrolled or symptomatic angina;
2. Myocardial infarction less than 6 months from study entry;
3. A history of arrhythmia requiring medication or clinically significant symptoms;
4. Uncontrolled or symptomatic congestive heart failure (> NYHA class 2);
5. Ejection fraction below the lower limit of the normal range. 6. severe infectious diseases (untreated tuberculosis, pulmonary aspergillosis).

7) Those deemed unsuitable for enrollment by the investigator

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | up to 12 months
  which evaluates the efficacy of patient induction therapy, including complete remission (CR), complete remission with incomplete blood count recovery (CRi), and morphologic leukemia-free state (MLFS)

SECONDARY OUTCOMES:
Minimal residual disease (MRD) | up to 12 months
  MRD percentage
overall survival (OS) | up to 12 months
  Overall Survival (OS) is used to evaluate all patients enrolled in a clinical trial, from the date of enrollment until death from any cause or the date of last follow-up for surviving patients.
relapse-free survival (RFS) | up to 12 months
  Relapse-Free Survival (RFS) is only used to evaluate patients who achieve complete remission (CR) through reinduction therapy. RFS is defined as the time from achievement of CR until death from any cause, relapse, or the date of last follow-up.
30-day mortality rate | Within 30 days after starting the medication
  The 30-day mortality rate is used to evaluate all patients enrolled in a clinical trial, and is defined as the percentage of patients who die within 30 days of starting chemotherapy.
adverse drug reactions | up to 12 months
  Adverse drug reactions during chemotherapy and follow-up

CONTACTS AND LOCATIONS:
Overall Officials: ZePing Zhou, Study Chair — The Second Affiliated Hospital of Kunming Medical University
Locations (1):
- The Second Affiliated Hospital of Kunming Medical University., Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dohner H, Weisdorf DJ, Bloomfield CD. Acute Myeloid Leukemia. N Engl J Med. 2015 Sep 17;373(12):1136-52. doi: 10.1056/NEJMra1406184. No abstract available. PMID 26376137
- [Background] Del Poeta G, Venditti A, Del Principe MI, Maurillo L, Buccisano F, Tamburini A, Cox MC, Franchi A, Bruno A, Mazzone C, Panetta P, Suppo G, Masi M, Amadori S. Amount of spontaneous apoptosis detected by Bax/Bcl-2 ratio predicts outcome in acute myeloid leukemia (AML). Blood. 2003 Mar 15;101(6):2125-31. doi: 10.1182/blood-2002-06-1714. Epub 2002 Nov 7. PMID 12424199
- [Background] Mei M, Aldoss I, Marcucci G, Pullarkat V. Hypomethylating agents in combination with venetoclax for acute myeloid leukemia: Update on clinical trial data and practical considerations for use. Am J Hematol. 2019 Mar;94(3):358-362. doi: 10.1002/ajh.25369. Epub 2018 Dec 13. PMID 30499168
- [Background] DiNardo CD, Jonas BA, Pullarkat V, Thirman MJ, Garcia JS, Wei AH, Konopleva M, Dohner H, Letai A, Fenaux P, Koller E, Havelange V, Leber B, Esteve J, Wang J, Pejsa V, Hajek R, Porkka K, Illes A, Lavie D, Lemoli RM, Yamamoto K, Yoon SS, Jang JH, Yeh SP, Turgut M, Hong WJ, Zhou Y, Potluri J, Pratz KW. Azacitidine and Venetoclax in Previously Untreated Acute Myeloid Leukemia. N Engl J Med. 2020 Aug 13;383(7):617-629. doi: 10.1056/NEJMoa2012971. PMID 32786187
- [Background] Wei AH, Strickland SA Jr, Hou JZ, Fiedler W, Lin TL, Walter RB, Enjeti A, Tiong IS, Savona M, Lee S, Chyla B, Popovic R, Salem AH, Agarwal S, Xu T, Fakouhi KM, Humerickhouse R, Hong WJ, Hayslip J, Roboz GJ. Venetoclax Combined With Low-Dose Cytarabine for Previously Untreated Patients With Acute Myeloid Leukemia: Results From a Phase Ib/II Study. J Clin Oncol. 2019 May 20;37(15):1277-1284. doi: 10.1200/JCO.18.01600. Epub 2019 Mar 20. PMID 30892988
- [Background] DiNardo CD, Maiti A, Rausch CR, Pemmaraju N, Naqvi K, Daver NG, Kadia TM, Borthakur G, Ohanian M, Alvarado Y, Issa GC, Montalban-Bravo G, Short NJ, Yilmaz M, Bose P, Jabbour EJ, Takahashi K, Burger JA, Garcia-Manero G, Jain N, Kornblau SM, Thompson PA, Estrov Z, Masarova L, Sasaki K, Verstovsek S, Ferrajoli A, Weirda WG, Wang SA, Konoplev S, Chen Z, Pierce SA, Ning J, Qiao W, Ravandi F, Andreeff M, Welch JS, Kantarjian HM, Konopleva MY. 10-day decitabine with venetoclax for newly diagnosed intensive chemotherapy ineligible, and relapsed or refractory acute myeloid leukaemia: a single-centre, phase 2 trial. Lancet Haematol. 2020 Oct;7(10):e724-e736. doi: 10.1016/S2352-3026(20)30210-6. Epub 2020 Sep 5. PMID 32896301
- [Background] DiNardo CD, Lachowiez CA, Takahashi K, Loghavi S, Xiao L, Kadia T, Daver N, Adeoti M, Short NJ, Sasaki K, Wang S, Borthakur G, Issa G, Maiti A, Alvarado Y, Pemmaraju N, Montalban Bravo G, Masarova L, Yilmaz M, Jain N, Andreeff M, Jabbour E, Garcia-Manero G, Kornblau S, Ravandi F, Konopleva MY, Kantarjian HM. Venetoclax Combined With FLAG-IDA Induction and Consolidation in Newly Diagnosed and Relapsed or Refractory Acute Myeloid Leukemia. J Clin Oncol. 2021 Sep 1;39(25):2768-2778. doi: 10.1200/JCO.20.03736. Epub 2021 May 27. PMID 34043428
- [Background] Wei H, Wang Y, Gale RP, Lin D, Zhou C, Liu B, Qiu S, Gu R, Li Y, Zhao X, Wei S, Gong B, Liu K, Gong X, Liu Y, Zhang G, Song Z, Wang Y, Li W, Mi Y, Wang J. Randomized Trial of Intermediate-dose Cytarabine in Induction and Consolidation Therapy in Adults with Acute Myeloid Leukemia. Clin Cancer Res. 2020 Jul 1;26(13):3154-3161. doi: 10.1158/1078-0432.CCR-19-3433. Epub 2020 Feb 6. PMID 32029439